CLINICAL TRIAL: NCT04154059
Title: Effects of a Strengthening Program for Foot-ankle Muscles in Clinical Aspects and Gait Biomechanics of People With Knee Osteoarthritis: a Randomized Blinded Clinical Trial
Brief Title: Strengthening Program for Foot-ankle Muscles in People With Knee Osteoarthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment of potential participants is suspended due to the covid-19 pandemic.
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Glauko André de Figueiredo Dantas, Principal Investigator (MSc), Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LabPlastUFSCar
Record Dates: First submitted 2019-10-31; First posted 2019-11-06 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
Keywords: Rehabilitation; Arthrosis; Therapeutic exercises; Feet
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients will receive a physical therapy intervention three times per week, for 8 weeks.
  Interventions: Other: Intervention Group
- Control Group (No Intervention): Patients will not receive any exercise treatment but they will keep their recommended clinical treatment.

INTERVENTIONS:
Other: Intervention Group — Patients will receive a physical therapy intervention for strengthening, stretching and functional training of ankle and foot.
  Other Names: Foot and ankle kinesiotherapy
  Arms: Intervention Group

SUMMARY:
The main objective of this trial is To evaluate the effect of an ankle and foot muscle strengthening program on pain, analgesic consumption, functionality, and lower limb biomechanics during gait in individuals with knee osteoarthritis.

DETAILED DESCRIPTION:
A randomized controlled trial will be performed with 76 patients with knee osteoarthritis. The participants will be randomly assigned into either a control group (no exercises; they will keep their recommended clinical treatment) or an intervention group which will receive 8-week physical therapy exercises, three times per week, under the supervision of a physiotherapist. Every exercise has its own progression depending on the subjects' execution, increasing in intensity and difficulty.

The subjects will be evaluated in 3 different moments (Baseline, immediately after treatment and 8 weeks follow-up).

The hypothesis of this study is that the intervention group will decrease pain and medication intake, and improve functional performance, increase isometric strength of the feet and production of beneficial biomechanical changes during walking compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis (KOA) based on clinical and radiological criteria of American College of Reumathology;
* KOA (Grade II and III - Radiological classification of Kellgreen and Laurence) in medial compartment of knee;
* Knee pain between 30 and 80 on the visual analogue scale;
* BMI < 35 kg/m2.

Exclusion Criteria:

* KOA isolated (Grade II and III - Radiological classification of Kellgreen and Laurence) in lateral compartment of knee;
* Lower limb strength training (3 times per week);
* Wear minimalist shoes for at least 6 hours a day and 5 days a week;
* Physical therapy in the previous 3 months;
* Having received steroid injections and hyaluronic acid intra-articular knee in previous periods of three and six months respectively;
* Previous history of surgery on knees, ankles and hips in the last 2 years;
* Neurological disease;
* Inflammatory arthritis (eg. rheumatoid arthritis);
* Asymptomatic OA of one or both knees.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline The WOMAC (Western Ontario and McMaster Universities) Pain Subscale at 8 and 16 weeks. | Baseline, 8 weeks and 16 weeks.
  The WOMAC pain subscale consists of five questions (Likert Scale) relating to the patient's pain in everyday situations. The Likert Scale version used for all WOMAC items are: none, mild, moderate, severe, and extreme. The sum of all items of pain subscale ranges from 0 to 20. Higher scores indicate worse pain.

SECONDARY OUTCOMES:
Change from baseline WOMAC (Western Ontario and McMaster Universities) Stiffness Subscale at 8 and 16 weeks. | Baseline, 8 weeks and 16 weeks.
  The stiffness subscale included in the WOMAC index consists of two questions (Likert Scale) relating articular function of the patient. The Likert Scale version used for all WOMAC items are: none, mild, moderate, severe, and extreme. The sum of all items of the stiffness subscale ranges from 0 to 8. Higher scores on the stiffness WOMAC subscale indicate worse articular function.
Change from baseline WOMAC (Western Ontario and McMaster Universities) Physical Function Subscale at 8 and 16 weeks. | Baseline, 8 weeks and 16 weeks.
  he physical function subscale included in the WOMAC index consists of seventeen questions (Likert Scale) relating to the patient's physical activities, or skills to move out and take care of themselves. The Likert Scale version used for all WOMAC items are: none, mild, moderate, severe, and extreme. The sum of all items of physical function subscale ranges from 0 to 68. Higher scores on the physical function WOMAC subscale indicate worse functional limitations.
Change from baseline WOMAC (Western Ontario and McMaster Universities) Total Score at 8 and 16 weeks | Baseline, 8 weeks and 16 weeks.
  The WOMAC total score is the sum of all subscale (pain, function and stiffness) (Likert Scale) relating to the patient's physical activities, or skills to move out and take care of themselves. The Likert Scale version used for all WOMAC items are: none, mild, moderate, severe, and extreme.
30-second Chair Stand Test | Baseline, 8 weeks and 16 weeks.
  The maximum number of chair stand repetitions possible in a 30 second period.
9-step Stair Climb Test | Baseline, 8 weeks and 16 weeks.
  The time (in seconds) it takes to ascend and descend a flight of stairs. Where possible, the 9-step stair test with 20cm (8 inch) step height and handrail is recommended.
40m (4x10m) Fast Paced Walk Test | Baseline, 8 weeks and 16 weeks.
  A test of walking speed over short distances and changing direction during walking. A fast-paced walking test that is timed over 4 x 10m for a total 40 m (convert time to speed).
Foot strength | Baseline, 8 weeks and 16 weeks.
  Hallux and lesser toes force measured by a pressure plate
Foot Kinematics during gait | Baseline, 8 weeks and 16 weeks.
  Foot joints and plantar arch motion during gait.The kinematics outcomes will be evaluate by mean inverse dynamics approach. To this procedure, we will use the kinematics data of the lower limbs assessed with six infrared cameras and the ground reaction force evaluated by mean a force platform.
Knee joint moments during gait | Baseline, 8 weeks and 16 weeks.
  Peak joint moment by inverse dynamic calculations. To this procedure, we will use the kinematics and kinetics data of the lower limbs assessed with six infrared cameras and the ground reaction force evaluated by mean a force platform.
Global Rating of Change Scale | 8 weeks and 16 weeks.
  GRCS assesses the clinical change perceived by the patient by comparing the onset of symptoms before and after treatment. "With respect to your knee injury, how do you describe your situation now compared to the start of treatment?" This numerical scale consists of 11 points (from -5 to +5: -5, extremely worse; 0, unchanged; +5, fully recovered). Higher scores indicate better recovery from the condition.
Paracetamol intake | Baseline, 8 weeks and 16 weeks.
  Paracetamol intake (500 mg), number of tablets per month.

CONTACTS AND LOCATIONS:
Locations (1):
- Glauko Dantas, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All data collected during the trial will be compiled electronically. Data integrity and validity will be verified at the time of data entry (edit checks). The project manager and research assistant will regularly monitor the study datasets and make recommendations regarding necessary protocol modifications or termination of all or part of the study. Participant data that underlie the results reported in this paper will be shared after blinding (text, tables, figures, appendices), immediately following publication. In addition, the study protocol and clinical trial report (both with the planned statistical analysis) will be made available by the researchers who proposed the methodology. Requests for data or any form of analysis should be directed to glauko.ft.andre@hotmail.com or tania@ufscar.br. Requesters will be asked to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Participant data that underlie the results reported in this paper will be shared after blinding (text, tables, figures, appendices), immediately following publication.
Access Criteria: Requests for data or any form of analysis should be directed to glauko.ft.andre@hotmail.com or tania@ufscar.br. Requesters will be asked to sign a data access agreement.

REFERENCES:
- [Result] Dantas G, Sacco ICN, Dos Santos AF, Watari R, Matias AB, Serrao PRMS, Pott-Junior H, Salvini TF. Effects of a foot-ankle strengthening programme on clinical aspects and gait biomechanics in people with knee osteoarthritis: protocol for a randomised controlled trial. BMJ Open. 2020 Sep 25;10(9):e039279. doi: 10.1136/bmjopen-2020-039279. PMID 32978204
- [Result] Dantas GAF, Sacco ICN, Ferrari AV, Matias AB, Watari R, Oliveira LVM, Marcon TR, Fatore JA, Pott-Junior H, Salvini TF. Effects of a foot-ankle muscle strengthening program on pain and function in individuals with knee osteoarthritis: a randomized controlled trial. Braz J Phys Ther. 2023 Jul-Aug;27(4):100531. doi: 10.1016/j.bjpt.2023.100531. Epub 2023 Aug 11. PMID 37603935